CLINICAL TRIAL: NCT01869816
Title: Implications of C1q/TNF-related Protein-3(CTRP-3) and Progranulin in Patients With Acutecoronary Syndrome and Stable Angina Pectoris
Brief Title: CTRP3 and Progranulin in Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: CAD(CTRP3,PRGL)
Record Dates: First submitted 2013-06-02; First posted 2013-06-05 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease
Keywords: CTRP-3; progranulin; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Acute coronary syndrome (ACS): Who were admitted to the coronary care units of the division of cardiology at Guro hospital in Korea University Medical Center. They have Acute myocardial infarction or unstable angina.
- Stable angina pectoris (SAP): Who were admitted to the coronary care units of the division of cardiology at Guro hospital in Korea University Medical Center. They have Stable angina.
- Control: Who were recruited from the participants for a routine health check-up in the Health Promotion Center of Korea University Guro Hospital.

SUMMARY:
Visceral obesity is the one of the major causes of cardiovascular morbidity and mortality in industrialized countries. Adipose tissue secretes various kinds of bioactive molecules termed adipokines which contribute to the development of obesity-related disorders including cardiovascular disease (CVD). Progranulin and CTRP3 are recently discovered novel adipokines. Therefore, the investigators tried to compare circulating CTRP-3 and progranulin levels in patients with CAD and investigated whether CTRP-3 or progranulin is significantly associated with CAD prevalence after adjustment for well-known CAD risk factors.

DETAILED DESCRIPTION:
CTRP-3 (synonyms CORS-26, cartducin and cartonectin) is a potent anti-inflammatory adipokine that inhibits proinflammatory pathways in monocytes and adipocytes. Using a recently developed enzymelinked immunosorbent assay (ELISA), we reported that circulating CTRP-3 levels were elevated in patients with glucose metabolism dysregulation.

Progranulin was identified as a key adipokine mediating high fat diet-induced insulin resistance and obesity through interleukin-6 (IL-6) in adipose tissue. We previously reported that progranulin levels were significantly higher in individuals with type 2 diabetes and were associated with macrophage infiltration in omental adipose tissue. Moreover, the expression of progranulin reduces inflammation and its degradation into granulins peptides enhances inflammation in atherosclerotic plaque, which may contribute to the progression of atherosclerosis There has been no previous report on the implication of CTRP-3 or progranulin in humans with cardiovascular disease (CAD). In the present study, we compared circulating CTRP-3 and progranulin levels in patients with CAD and investigated whether CTRP-3 or progranulin is significantly associated with CAD prevalence after adjustment for well known CAD risk factors.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction
* unstable angina
* stable angina pectoris

Exclusion Criteria:

For control group, we exclude the participants who had

* a history of CVD (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* type 2 diabetes
* stage 2 hypertension (resting blood pressure, ≥160/100 mmHg)
* malignancy
* severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome (ACS) patients, who were admitted to the coronary care units of the Division of Cardiology at Guro Hospital in Korea University Medical Center.
  Control subjects were recruited from the participants for a routine health check-up in the Health Promotion Center of Korea University Guro Hospital.
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2011-03-01; Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
CTRP3 | 16 months
  CTRP3 (ng/ml)

SECONDARY OUTCOMES:
SBP | 16 months
  SBP (mmHg)
LDL cholesterol | 16 months
  LDL (mg/dl)
hsCRP | 16 months
  hsCRP (mg/dl)
creatinine | 16 months
  creatinine (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, M.D., Principal Investigator — Korea University
Locations (1):
- Korea University Guro Hospital Dept. of Endocrinology, Seoul, South Korea